CLINICAL TRIAL: NCT02431793
Title: EHR-Based Medication Complete Communication Strategy to Promote Safe Opioid Use
Acronym: EMC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Danielle McCarthy, Assistant Professor in Emergency Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HS023459-01 (AHRQ)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Opioid Use, Unspecified
Keywords: Opioids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (No Intervention): Employ the standard of care, no intervention
- EMC2 strategy (Experimental): Patients of providers randomized to EMC2 arm will received educational tool from the ED to support the understanding and safe use of opioids.
  1. A single-page medication information sheet with content from a patients perspective and following health literacy best practices.
  2. Prescribing instructions will be adapted to the Universal Medication Scheduled Take-Wait-Stop regimen for both the prescribing and dispensing of the medicine. This format uses simplified text and numeric characters to detail dose.
  3. Provider counseling prompts: The providers for patients in this arm will be prompted to encourage counseling both in the ED and at follow-up time points. These prompts include: 1) An automated prompt to the ED physician upon signing the order; 2) an automated message to the PCP (if an in-system PCP) notifying them of the ED visit, new prescription, and counseling request; and 3) a request for the pharmacist to counsel patient printed automatically on the prescription.
  Interventions: Behavioral: EMC2 Strategy
- EMC2 strategy + SMS Text Reminders (Experimental): In addition to the EMC2 Strategy Arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
  Interventions: Behavioral: EMC2 Strategy; Behavioral: SMS Text Reminders

INTERVENTIONS:
Behavioral: EMC2 Strategy — Patients of providers randomized to the EMC2 arm will received study related educational tools at the time of their discharge including: (a) health-literacy appropriate MedSheet for hydrocodone-acetaminophen and (b) prescription written with Universal Medication Schedule Take-Wait-Stop language. Additionally, providers related to the patient will be prompted to counseling the patient including: (c) (c-1) ED providers prompted via EHR, (c-2) PCP prompted to counsel on follow-up visit via automated message and (c-3) pharmacists prompted to counsel via request printed on prescription.
  Arms: EMC2 strategy; EMC2 strategy + SMS Text Reminders
Behavioral: SMS Text Reminders — In addition to the components of the EMC2 strategy arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
  Arms: EMC2 strategy + SMS Text Reminders

SUMMARY:
The purpose of this study is to test the effectiveness of an electronic health record based strategy in promoting safe use of opioid medications after an Emergency Department (ED) visit. The electronic health record (EHR)-based strategy was designed to enhance provider counseling about opioids and to standardize and simplify the information that patients receive.

DETAILED DESCRIPTION:
Research has shown that patients frequently leave the emergency department without sufficient knowledge about how to safely use their newly prescribed opioid pain relievers. Additionally, educational interventions have the ability to increase patient knowledge about medications. In this study, education interventions will be implemented at the level of the EHR and prompt increased provider counseling with a goal of improving patient knowledge and safe use of opioids after ED discharge.

The investigators will conduct a three-arm provider randomized controlled trial among English-speaking adults prescribed hydrocodone-acetaminophen to evaluate the effectiveness of the EMC2 strategy, with and without Short Message Service (SMS) text reminders, to improve patient understanding and safe use of their medication compared to usual care. This study will be conducted at an urban, academic emergency department (annual volume >85,000 patient visits) in Chicago, Illinois. English speaking patients will be recruited and assessed in person at baseline, and by phone at 2-4 days, 7-14 days, and 1 month after recruitment.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to enroll and remain in the study, patient subjects must meet all of the following criteria:

  1. Patient age 18 years and older
  2. English language speaking
  3. prescribed pill form of hydrocodone-acetaminophen opioid pain reliever
  4. own a cell phone with text messaging capabilities
  5. the patient is the person primarily responsible for administering medication

Exclusion Criteria:

* Subjects will be excluded from the study if any of the following conditions are met:

  1. Aged <18
  2. non-English speaking
  3. clinically unstable, psychologically impaired or intoxicated as judged by research staff member or emergency physician
  4. chronic opioid use, defined as daily or near daily use of opioid pain relievers for the past 90 days
  5. admitted to hospital
  6. unable to complete follow up phone interviews
  7. pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle McCarthy, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] McCarthy DM, Kim HS, Hur SI, Lank PM, Arroyo C, Opsasnick LA, Piserchia K, Curtis LM, Wolf MS, Courtney DM. Patient-Reported Opioid Pill Consumption After an ED Visit: How Many Pills Are People Using? Pain Med. 2021 Feb 23;22(2):292-302. doi: 10.1093/pm/pnaa048. PMID 32219431
- [Derived] McCarthy DM, Curtis LM, Courtney DM, Cameron KA, Lank PM, Kim HS, Opsasnick LA, Lyden AE, Gravenor SJ, Russell AM, Eifler MR, Hur SI, Rowland ME, Walton SM, Montague E, Kim KA, Wolf MS. A Multifaceted Intervention to Improve Patient Knowledge and Safe Use of Opioids: Results of the ED EMC2 Randomized Controlled Trial. Acad Emerg Med. 2019 Dec;26(12):1311-1325. doi: 10.1111/acem.13860. Epub 2019 Nov 19. PMID 31742823
- [Derived] Neill LA, Kim HS, Cameron KA, Lank PM, Patel DA, Hur SI, Opsasnick LA, Curtis LM, Eifler MR, Courtney DM, Wolf MS, McCarthy DM. Who Is Keeping Their Unused Opioids and Why? Pain Med. 2020 Jan 1;21(1):84-91. doi: 10.1093/pm/pnz025. PMID 30903661
- [Derived] McCarthy DM, Courtney DM, Lank PM, Cameron KA, Russell AM, Curtis LM, Kim KA, Walton SM, Montague E, Lyden AL, Gravenor SJ, Wolf MS. Electronic medication complete communication strategy for opioid prescriptions in the emergency department: Rationale and design for a three-arm provider randomized trial. Contemp Clin Trials. 2017 Aug;59:22-29. doi: 10.1016/j.cct.2017.05.003. Epub 2017 May 4. PMID 28479220

RESULTS

PARTICIPANT FLOW:
Groups:
- EMC2 Strategy: Patients of providers randomized to EMC2 arm will receive educational tool from the Emergency Department (ED) to support the understanding and safe use of opioids.
  1. A single-page medication information sheet with content from a patients perspective, following health literacy best practices.
  2. Prescribing instructions will be adapted to the Universal Medication Scheduled Take-Wait-Stop regimen for both prescribing and dispensing of the medicine. This format uses simplified text and numeric characters to detail dose.
  3. Provider counseling prompts: The providers for patients in this arm will be prompted to encourage counseling both in the ED and at follow-up time points. These prompts include: 1) An automated prompt to the ED physician upon signing the order; 2) an automated message to the PCP (if in-system PCP) notifying them of ED visit, new prescription, and counseling request; and 3) a request for the pharmacist to counsel patient printed automatically on the prescription.
- EMC2 Strategy + SMS Text Reminders: In addition to the EMC2 Strategy Arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
  EMC2 Strategy: Patients of providers randomized to the EMC2 arm will received study related educational tools at the time of their discharge including: (a) a single-page medication information sheet for hydrocodone-acetaminophen and (b) prescription written with Universal Medication Schedule Take-Wait-Stop language. Additionally, providers related to the patient will be prompted to counseling the patient including: (c) (c-1) ED providers prompted via electronic health record (EHR), (c-2) PCP prompted to counsel on follow-up visit via automated message and (c-3) pharmacists prompted to counsel via request printed on prescription.
  SMS Text Reminders: In addition to the components of the EMC2 strategy arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
Period: Overall Study
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Started | 202 | 243 | 207
Completed T1 (3-5 Days Post Enrollment) | 136 | 180 | 143
Completed T2 (7-14 Days Post Enrollment) | 95 | 141 | 107
Completed T3 (30 Days Post Enrollment) | 85 | 113 | 93
Completed | 83 | 109 | 90
Not Completed | 119 | 134 | 117
Not completed — Ineligible doe to not filling Rx | 11 | 7 | 8
Not completed — Withdrawal by Subject | 7 | 5 | 5
Not completed — Lost to Follow-up | 101 | 122 | 104

BASELINE CHARACTERISTICS:
Groups:
- EMC2 Strategy: Patients of providers randomized to EMC2 arm will received educational tool from the ED to support the understanding and safe use of opioids.
  1. A single-page medication information sheet with content from a patients perspective and following health literacy best practices.
  2. Prescribing instructions will be adapted to the Universal Medication Scheduled Take-Wait-Stop regimen for both the prescribing and dispensing of the medicine. This format uses simplified text and numeric characters to detail dose.
  3. Provider counseling prompts: The providers for patients in this arm will be prompted to encourage counseling both in the ED and at follow-up time points. These prompts include: 1) An automated prompt to the ED physician upon signing the order; 2) an automated message to the PCP (if an in-system PCP) notifying them of the ED visit, new prescription, and counseling request; and 3) a request for the pharmacist to counsel patient printed on the prescription.
- EMC2 Strategy + SMS Text Reminders: In addition to the EMC2 Strategy Arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
  EMC2 Strategy: Patients of providers randomized to the EMC2 arm will received study related educational tools at the time of their discharge including: (a) health-literacy appropriate MedSheet for hydrocodone-acetaminophen and (b) prescription written with Universal Medication Schedule Take-Wait-Stop language. Additionally, providers related to the patient will be prompted to counseling the patient including: (c) (c-1) ED providers prompted via EHR, (c-2) PCP prompted to counsel on follow-up visit via automated message and (c-3) pharmacists prompted to counsel via request printed on prescription.
  Short Message Service (SMS) Text Reminders: In addition to the components of the EMC2 strategy arm, patients will received daily text message reminders about the safe use of opioids for 7 days.
- Total: Total of all reporting groups
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders | Total
Number analyzed (Participants) | 202 | 243 | 207 | 652
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.2) | 42.3 (14.4) | 41.3 (13.3) | 42.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 135 | 124 | 372
  Male | 89 | 108 | 83 | 280
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Two individuals refused to identify their race, so the total population analyzed for race was 650 as opposed to 652.
  Participants
    Race: number analyzed (Participants) | 201 | 242 | 207 | 650
    Race: White | 95 | 110 | 100 | 305
    Race: African American | 66 | 71 | 63 | 200
    Race: Other | 40 | 61 | 44 | 145
Health Literacy (NVS) [Count of Participants; unit: Participants]
  Limited/Marginal Literacy | 71 | 80 | 68 | 219
  Adequate Literacy | 131 | 163 | 139 | 433
Income [Count of Participants; unit: Participants] — Population: 70 individuals refused to/felt uncomfortable identifying their income, so the total population analyzed for income was 582 as opposed to 652.
  Participants
    number analyzed (Participants) | 184 | 223 | 175 | 582
    < $40,000 | 60 | 69 | 49 | 178
    $40,000-$100,000 | 68 | 78 | 56 | 202
    >$100,000 | 56 | 76 | 70 | 202

OUTCOME MEASURES:

1. Primary Outcome: Safe Medication Dosing (Prescription Understanding)
Description: Patient's ability to demonstrate correctly dosing their prescription opioid-acetaminophen pain reliever will be assessed through a series of questions. Correct dosing will be scored for each medication as yes/no reflecting having demonstrated all of the following: proper dose (# of pills), appropriate spacing (hours between doses), and total daily dose (not exceeding recommended daily dose).
Time Frame: 7-14 days after enrollment
Population: The population for this analysis includes anyone who completed the demonstrated dosing task at T2 (7-14 days post enrollment). The reported results represent the predicted probability of correctly demonstrating dosing, adjusting for health literacy and physician inter-correlation.
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Number analyzed (Participants) | 77 | 107 | 86
probability | 0.67 [0.55 to 0.77] | 0.83 [0.75 to 0.89] | 0.79 [0.69 to 0.87]

2. Secondary Outcome: Medication Knowledge
Description: The identification of the medications purpose, side effects, risks, warnings and benefits will be assessed through a structured questionnaire. Patients will be asked about each of the above via structured, open-ended items. Additionally, select questions from the validated Patient Opioid Education Measure and patient satisfaction questions will be included. The Patient Knowledge Score was developed from these questions, with a score range of 0 to 10. A higher score on the scale represents better patient knowledge.
Time Frame: 7-14 days after enrollment
Population: The population for this analysis includes anyone who answered the knowledge questions at T2 (7-14 days post enrollment). The reported results represent the mean knowledge score (0-10), adjusting for health literacy, income, race and physician inter-correlation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Number analyzed (Participants) | 73 | 113 | 125
score on a scale | 5.48 [5.13 to 5.84] | 5.46 [5.16 to 5.75] | 6.06 [5.71 to 6.41]

3. Secondary Outcome: Proper Medication Use (Medication Diary)
Description: Patients medication use will be assessed through a combination of a home medication diary (collected at 7-14 days post enrollment), pill count, and patient report of medication use.
Time Frame: 10 day medication diary
Population: The population for this analysis includes anyone who returned their medication diary with medication information filled out. The reported results represent the predicted probability of correctly using medication (without errors), adjusting for physician inter-correlation.
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Number analyzed (Participants) | 75 | 98 | 85
probability | 0.52 [0.40 to 0.63] | 0.66 [0.56 to 0.75] | 0.65 [0.54 to 0.75]

4. Secondary Outcome: Current Opioid Misuse Measure (COMM)
Description: Select questions from the Current Opioid Misuse Measure (COMM) will be used to assess if patients are safely taking their prescription opioids.
Time Frame: 7-14 days after enrollment
Population: The population for this analysis includes anyone who answered select COMM questions at T2 (7-14 days post enrollment). The reported results represent those who safely took their opioid medications, adjusting for health literacy, income, race and physician inter-correlation.
Measure: Least Squares Mean (95% Confidence Interval); unit: probability
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Number analyzed (Participants) | 90 | 131 | 90
probability | 0.70 [0.58 to 0.79] | 0.78 [0.70 to 0.85] | 0.71 [0.60 to 0.81]

5. Secondary Outcome: Pain Score
Description: Pain scores through structured questions about use in the past 24 hours were collected from participants. Pain Score was assessed on a scale from 0 to 10, where higher numbers represent higher pain scores.
Time Frame: 7-14 days after enrollment
Population: The population for this analysis includes anyone who answered the pain score questions at T2 (7-14 days post enrollment). The reported results represent the mean pain score (0-10), adjusting for health literacy, income, race and physician inter-correlation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
Number analyzed (Participants) | 88 | 116 | 75
score on a scale | 2.76 [2.21 to 3.31] | 2.47 [2.01 to 2.94] | 2.60 [2.03 to 3.17]

ADVERSE EVENTS:
Time Frame: 30 day
Description: revisit resulting in admission or ICU care related to their prescribed opioid/acetaminophen (acetaminophen overdose, opioid overdose)
Arm/Group | Usual Care | EMC2 Strategy | EMC2 Strategy + SMS Text Reminders
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/243 | 0/207
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/243 | 0/207
Other Adverse Events (participants affected / at risk) | 0/202 | 0/243 | 0/207

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT02431793/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02431793/SAP_001.pdf